CLINICAL TRIAL: NCT00963729
Title: A Neoadjuvant Study of Chemotherapy Versus Endocrine Therapy in Postmenopausal Patients With Primary Breast Cancer
Brief Title: Chemotherapy or Letrozole Before Surgery in Treating Postmenopausal Women With Breast Cancer That Can Be Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: ICCRU-NEOcent-C-21-07; CDR0000641383 (Registry Identifier: PDQ (Physician Data Query)); ICCRU-NEOcent-C-21-07; EU-20936; EUDRACT-2006-003596-12; ISRCTN77234840
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: estrogen receptor-positive breast cancer; recurrent breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Epirubicin; Fluorouracil; Letrozole

ARMS (2):
- Arm I (Experimental): Patients receive fluorouracil IV, epirubicin IV, and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cyclophosphamide; Drug: docetaxel; Drug: epirubicin hydrochloride; Drug: fluorouracil
- Arm II (Experimental): Patients receive oral letrozole daily for 18-23 weeks until day of surgery.
  Interventions: Drug: letrozole

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Arms: Arm I
Drug: docetaxel — Given IV
  Arms: Arm I
Drug: epirubicin hydrochloride — Given IV
  Arms: Arm I
Drug: fluorouracil — Given IV
  Arms: Arm I
Drug: letrozole — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by reducing the production of estrogen. It is not yet known whether giving more than one drug (combination chemotherapy) or giving letrozole before surgery is more effective in treating women with breast cancer.

PURPOSE: This randomized phase III trial is studying giving combination chemotherapy before surgery to see how well it works compared with letrozole given before surgery in treating postmenopausal women with breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare the efficacy and tolerability of cytotoxic chemotherapy versus aromatase inhibition for the down-staging of strongly ER+ primary breast cancer in postmenopausal women.
* To identify biological predictors of response to these two treatment modalities.

OUTLINE: This is a multicenter pilot, feasibility study followed by a randomized study. In the pilot study, a record of all patients screened and invited to participate in the study is compiled. Reasons for failure to recruit will be recorded. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive fluorouracil IV, epirubicin IV, and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients who do not achieve at least partial response after 3 courses receive docetaxel IV on day 1 of 3-week courses for an additional 3 courses.
* Arm II: Patients receive oral letrozole daily for 18-23 weeks until day of surgery.

Patients in both arms undergo surgery at week 18-23. Most patients then receive adjuvant therapy.

Quality of life is assessed at baseline, periodically during study treatment, and then during follow up.

Blood is collected pre-treatment, at mid-treatment, and before surgery. Blood is then collected every 6 months for 2 years. Blood samples and preserved tumor samples are used for correlative studies.

After completion of surgery, patients are followed up at least annually for 10 years.

PROJECTED ACCRUAL: A total of 40 patients for the pilot study and 716 patients for the phase III study will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven primary invasive breast cancer that is thought to be suitable for neoadjuvant treatment

  * No cytological proof of malignancy only
  * T2 tumor or greater (≥ 20 mm by ultrasound) or any T stage with nodal disease ≥ 20 mm diameter on ultrasound assessment
  * No evidence of distant metastatic disease as disclosed by bone scan, liver, and chest imaging
* Definite indication for neoadjuvant and adjuvant chemotherapy
* Primary tumor amenable to biopsy
* No inoperable disease that is judged very unlikely to be rendered operable by neoadjuvant treatment
* No inflammatory breast cancer
* No bilateral invasive breast cancer
* HER-2 positivity is NOT an exclusion criterion in the feasibility (pilot) study
* Estrogen receptor (ER) positive tumor

  * No ER-poor disease as defined locally (e.g., H-score < 100, Allred 3/4/5)
  * Allred 6/7/8, H-score H ≥100 allowed

PATIENT CHARACTERISTICS:

* Postmenopausal, meeting 1 of the following criteria:

  * Over 12 months since last menstrual period
  * Postmenopausal gonadotrophin levels (luteinizing hormone or follicle-stimulating hormone levels above local criteria)
  * Postmenopausal estradiol levels below local criteria
  * Prior bilateral oophorectomy
  * Menopause induced by gonadotrophin-releasing hormone not allowed
* WHO performance status 0 or 1
* WBC ≥ 3.0 × 10^9/L
* ANC ≥ 1.5 × 10^9/L
* Platelets ≥ 100 × 10^9/L
* Hemoglobin > 9 g/dL
* AST/ALT ≤ 1.5 times upper limit of normal (ULN)
* Serum bilirubin ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 1.5 times ULN
* Serum creatinine ≤ 1.5 times ULN
* No active, uncontrolled infection
* No malignancy within the past 10 years except for basal cell carcinoma or cervical carcinoma in situ

  * Treatment for previous malignancy confined to resection alone
* No concomitant medical, psychiatric, or geographic problems that might prevent completion of treatment or follow-up
* No known severe hypersensitivity to aromatase inhibitors
* No contraindication to receiving aromatase inhibitors (clinical evidence or recorded history of osteoporosis)
* No other serious illness or medical condition including any of the following:

  * Congestive heart failure or unstable angina pectoris
  * Myocardial infarction within the past year
  * Uncontrolled hypertension or high-risk uncontrolled arrhythmias
  * History of significant neurologic or psychiatric disorders, including psychotic disorders, dementia, or seizures, that would prohibit the understanding and giving of informed consent
  * Active peptic ulcer
  * Unstable diabetes mellitus
* No definite contraindications for the use of corticosteroids
* No contraindication to receiving combination anthracycline/taxane chemotherapy
* Willing to undergo repeat biopsies

PRIOR CONCURRENT THERAPY:

* No hormone replacement therapy within 4 weeks of starting treatment
* No chronic oral treatment with corticosteroids unless initiated > 6 months prior to study entry and at low dose (≤ 20 mg methylprednisolone or equivalent)
* No concurrent warfarin or heparin therapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Feasibility of patient recruitment (pilot)
Feasibility of tissue collection (pilot)
Ultrasound (or mammogram) response rate

SECONDARY OUTCOMES:
Clinical response rate
Radiologic response rate by ultrasound (pilot)
Quality of life
Pathological complete response rate (pCR) defined as no residual invasive or pre-invasive carcinoma in breast or axilla (pilot)
Plasma DNA changes in relation to treatment response
Rate of conservation surgery
Degree of pathological response
Ki-67 changes and its relationship to treatment response
Length of time to maximum response within the treatment period
Tolerability of the various treatments
Disease-free survival
Overall survival
MRI response

CONTACTS AND LOCATIONS:
Overall Officials: R. Charles Coombes, MD, MRCP, FRCP, PhD, FMedSci, Study Chair — Charing Cross Hospital
Locations (5):
- Asan Medical Center - University of Ulsan College of Medicine, Seoul, South Korea
- United Kingdom (4):
  - West Middlesex University Hospital, Isleworth, England
  - Guy's Hospital, London, England
  - St. Mary's Hospital, London, England
  - Charing Cross Hospital, London, England